CLINICAL TRIAL: NCT03276819
Title: A Clinical and Biological Umbrella Protocol for Smoker or Non-smoker Patients With Oral Potentially Malignant Lesions (OPML) or Head and Neck Squamous Cell Carcinoma (HNSCC) (IHNPACT UMBRELLA)
Brief Title: A Clinical and Biological Umbrella Protocol for Smoker or Non-smoker Patients With OPML or HNSCC
Acronym: UMBRELLA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination of the study, since July 31, 2020 for insufficient recruitment
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IHNPACT Umbrella
Record Dates: First submitted 2017-09-04; First posted 2017-09-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Premalignant Lesion; Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Oral potentially malignant lesions (OPML); Head and neck squamous cell carcinoma (HNSCC); Biomarkers; Smoking cessation program; Loss of heterozigoty (LOH); Medico-economics; Sociology; Psychology
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Tobacco Products; Ethanol

STUDY DESIGN:
Intervention Model Description: Cohort A : Patients with OPML Cohort B : Patients with resectable HNSCC requiring postoperative radiotherapy or chemoradiation and which are either current smokers motivated to quit or reformed smokers within 3 months before the diagnosis of a resectable HNSCC Cohort C : Patients with resectable HNSCC wich are not eligible to cohort B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Samples collection and Tobacco and alcohol status follow-up for patient with OPML:
  Follow-up of the lesions (pictures, biopsies, brushes), malignant transformation oversight, smoking and alcohol status follow-up (questionnaires), blood and saliva samples
  Interventions: Procedure: Samples collection; Behavioral: Tobacco and alcohol status follow-up
- Cohort B (Experimental): Samples collection; Psychological and Sociological evaluation; Intensive and sustained smoking cessation program; Tobacco and alcohol status follow-up for patient with resectable HNSCC requiring postoperative radiotherapy or chemoradiation and which are either current smokers motivated to quit or reformed smokers within 3 months before the diagnosis of a resectable HNSCC.
  Randomization 1:1, arm 1 = minimal tobacco cessation intervention, arm 2 = intensive and sustained smoking cessation program.
  Smoking and alcohol status follow-up, adhesion to the smoking cessation program, tumoral follow-up, second malignant lesion, tumoral collection, blood biomarkers research
  Interventions: Procedure: Samples collection; Behavioral: Psychological and Sociological evaluation; Behavioral: Intensive and sustained smoking cessation program; Behavioral: Tobacco and alcohol status follow-up
- Cohort C (Experimental): Samples collection and Tobacco and alcohol status follow-up for patients with resectable HNSCC wich are not eligible to cohort B Smoking and alcohol status follow-up (questionnaires), tumoral follow-up, second malignant lesion and OPML lesion appearance oversight, tumoral collection, blood biomarkers research
  Interventions: Procedure: Samples collection; Behavioral: Tobacco and alcohol status follow-up

INTERVENTIONS:
Procedure: Samples collection — OPML biopsy or resection, biopsy of normal oral mucosa, surgical specimen of HNSCC, saliva samples, buccal brushes, blood samples
Behavioral: Psychological and Sociological evaluation — Cohort B ....
  Arms: Cohort B
Behavioral: Intensive and sustained smoking cessation program — Evaluation of efficacy of the smoking cessation program (intensive and sustained versus minimal)
  Arms: Cohort B
Behavioral: Tobacco and alcohol status follow-up — Evaluation of the tobacco and alcohol status all along the study (questionnaires)

SUMMARY:
This is a multicenter minimal risk or burden prospective 3-cohort follow-up and monitoring study that aims to collect clinical, socio-psychological, medico-economics data and biospecimens for patients with oral potentially malignant lesions (OPML) or resectable head and neck squamous cell carcinoma (HNSCC) :

* Cohort A: OPML patients.
* Cohort B (specific design): smokers (adults who have smoked at least 100 cigarettes in their lifetime) motivated to quit - either current smokers (who currently smokes cigarettes every day (daily) or some days (nondaily)) or former smokers (adults who have smoked at least 100 cigarettes in their lifetime, but say they currently do not smoke) who stops smoking within 3 months prior to the diagnosis - with a resectable HNSCC requiring postoperative radiotherapy or chemoradiation.
* Cohort C: Patients with resectable HNSCC non-eligible to cohort B.

The primary objective of this study is the identification of biomarkers (predictive of malignant transformation or second primary tumor) and new strategies for prevention and therapy, mainly through extensive genomic, epigenomic and immune characterization of OPML and HNSCC.

DETAILED DESCRIPTION:
The long-term goal of this study is to reduce the incidence of HNSCC which may impact as well other smoking-related cancers. It may be interesting to foster excellent translational research towards the target of reducing the incidence of HNSCC by developing a global and personalized approach for prevention and treatment of HNSCC. The only way to reach this goal is to develop an ambitious program that coordinates the efforts of experts from various fields (surgeons, medical oncologists and addictologists, scientists, sociologists and economists) that will work together toward the same goal.

This study intends to gather a large scale clinical, sociological, psychological data gathering combined to a unique set of biospecimens collected prospectively including oral preneoplastic disease and resectable HNSCC. This represents a unique setting to develop multidisciplinary studies including a translational research component (validation and discovery of biomarkers, high throughput molecular studies to understand the dynamics of molecular changes and identify new strategies for prevention), a sociopsychological component and an addiction component that aim to increase the percentage of patients entering a process of weaning, as well as a medico-economics component that intend to evaluate the impact of new approaches that may emerge from our work.

In summary, this study proposes to prospectively collect clinical, sociopsychological, medico-economics data and biospecimens in patients included in 3 different cohorts. Cohort A will include patients with OPML, either from smokers/drinkers (S/D) or non-smokers/non-drinkers (NS/ND), while cohort B and C will include patients with HNSCC eligible to upfront surgical resection. Patients in cohort B will be included in an interventional randomized clinical trial evaluating an intensive and sustained smoking cessation program.

In patients with OPML, no standard workup and treatment plan is recommended. OPMLs biopsy is important to identify patients with high grade dysplasia and in situ carcinoma who should undergo surgical resection of the OMPLs if possible. Although LOH status in OPML biopsies or buccal brushes has been evaluated in this population as a biomarker of risk to develop oral cancer, it is not routinely performed. More studies are required to validate their value as a biomarker of risk in a prospective setting and to identify the best set of biomarkers. In smokers and/or excessive alcohol drinkers, it is critical to counsel and help patients quit and it should be part of the standard of care. Unfortunately, this is not always the case. Studies of chemopreventive agents have not resulted in the development of an intervention that can be considered as standard of care.

Despite the accumulated knowledge, no comprehensive molecular characterization of OPML is available. Identification of new targets for prevention and therapy, mainly with genomic, epigenomic and immune characterization of OPML is critical. Cohort A will allow to prospectively collect clinical information and biospecimens (biopsies, buccal brushes and saliva). These unique resources will allow to confirm the value of LOH as a biomarker of risk and develop standardized procedures for sample processing that can be transferred in the routine setting, validate or identify other biomarkers and improve risk assessments beyond LOH, to understand the spatial and temporal dynamics of molecular changes that may help predicting oral cancer risk, identify relevant targets and suggest new chemoprevention strategies including immunoprevention interventions. Furthermore, patients included in this cohort will benefit from standardized care plans and state of the art smoking and alcohol cessation programs according to current recommendations, and will be given the opportunity to participate in future chemoprevention studies that may be embedded in the near future in the umbrella protocol.

In patients with resectable HNSCC (cohorts B and C), smoking and alcohol cessation is one important step in the management. They allow reducing treatment-related morbidity and improving radiation and chemoradiation efficacy. It is tempting to believe that they may also improve patients' quality of life as in the general population, and reduce the risk of second primary tumor (SPT). Available data focusing on patients with HNSCC and smoking cessation is scarce. Although the diagnosis and treatment of patients with HNSCC favors smoking cessation, a significant proportion of former smokers are actively smoking during follow-up despite having completed treatments associated with substantial morbidity. The literature review shows that the range of patients that continue to smoke at one year is in the range of 21-41%. Of note, those smoking quit rates at one year are based on patient self-reporting without biological confirmation in the majority of the cases, which clearly overestimates quit rates. Smoking cessation programs currently available lead to disappointing results. HNSCC patients with smoking addiction harbor the highest risk of SPTs. In this vulnerable population, beyond early management of nicotine dependence, new strategies / innovative interventional approaches are warranted. Preliminary results from a monocentric study indicate that an active intervention in this challenging population may lead to encouraging results in motivated patients. Furthermore, an intensive smoking cessation program implemented during radiation therapy is feasible in this population of patients. In cohort B, the efficacy of an intensive and sustained smoking cessation program in a randomized cohort of these patients at highest risk with potentially curable HNSCC (cohort B) will be evaluated, with the hypothesis that an intensive and sustained smoking cessation program led by an addictologist or a tobacco treatment specialist (TTS) during radiation therapy may improve the 6- and 12-month quite-rate compared with a minimal tobacco cessation intervention. Among secondary objectives of this trial, medico-economics information will be gathered to provide an initial assessment of the cost-effectiveness of the experimental versus standard arms.

Cohort C will allow prospective collection of clinical information and biospecimens (biopsies, buccal brushes and saliva) only. Patients will benefit from state of the art smoking and alcohol cessation programs according to current recommendations.

Well-annotated cohorts of patients with HNSCC are scarce. Information and biospecimens collected in cohorts B and C will provide unique resources to identify biomarkers of risk of recurrence and SPT.

Having access to large scale information and to biospecimens in patients with preneoplastic disease (cohort A) who may or may not develop smoking/alcohol related cancers, and with HNSCC (cohorts B and C) who may develop disease recurrence or SPT, represent a unique opportunity to understand the dynamics of molecular changes and their interaction with smoking cessation and/or alcohol withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the day of consenting to the study (or at the day of randomization for cohort B patients not included in the global study)
2. Patients with OPML: at least one lesion ≥ 5 mm (Cohort A only)
3. Patients with surgically resectable HNSCC not treated with preoperative chemotherapy, pT1-4 N0-3 M0 (Cohort B only)
4. Patients with surgically resectable HNSCC not treated with preoperative chemotherapy and non-eligible to cohort B (Cohort C only)
5. PS ECOG ≤ 1
6. Treatment plan incorporating surgery and radiation therapy (or at the day of randomization for cohort B patients not included in the global study)
7. Smoker = Adult who have smoked at least 100 cigarettes in his/her lifetime (Cohort B only)
8. Current smoker (who currently smokes cigarettes every day (daily) or some days (nondaily)) or former smoker (who says he/she doesn't smoke) who stops smoking within 3 months prior to diagnosis (Cohort B only)
9. Motivation to quit smoking evaluated by the Richmond test (Cohort B only)
10. Without subordination motivation to quit smoking (Cohort B only)
11. Covered by a medical insurance
12. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment

Exclusion Criteria:

1. Non-stabilized cognitive disorder
2. Synchronous malignancy (Cohort A only)
3. History of malignant disease outside the upper aerodigestive tract, except skin carcinoma
4. Substance use disorder other than smoking (cigarette and cannabis) and alcohol (Cohort B only)
5. Use of nicotine replacement therapy, bupropion, varenicline on last 3 months (Cohort B only)
6. Undergoing on last 3 months' behavioral and cognitive therapy for smoking cessation (Cohort B only)
7. Patient included in a clinical trial evaluating interventions for smoking cessation (Cohort B only)
8. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
9. Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Biomarkers | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Prevalence of LOH and/or other candidate biomarkers in OPML and normal mucosa : study of their spatial and temporal dynamic changes and explore their association with the risk of developing oral cavity squamous cell carcinoma, recurrent disease or second primary tumor (blood samples, buccal biopsies, buccal cells)

SECONDARY OUTCOMES:
alcohol quit | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Evaluation of alcohol quit rates for addicted patients (cohorts A and C only)
smoking quit | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Evaluation of smoking quit rates for addicted patients (cohorts A and C only)
cannabis quit | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Evaluation of cannabis quit rates for addicted patients (cohorts A and C only)
Preclinical models of oral mucosa | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Patient-derived preclinical models of oral normal mucosa from smokers/drinkers and non smokers/non drinkers
Preclinical models of OPML | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Patient-derived preclinical models of OPML from smokers/drinkers and non smokers/non drinkers
Preclinical models of HNSCC | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 from inclusion
  Patient-derived preclinical models of HNSCC from smokers/drinkers and non smokers/non drinkers
Efficacy of intensive and sustained smoking cessation program | Month 6, Month 12 after randomization
  Evaluation of the efficacy of an experimental, intensive and sustained smoking cessation program, versus minimal tobacco cessation intervention, in helping patients with HNSCC to achieve long-term abstinence (at 12 months after randomization), middle term-abstinence (at least 6 months after randomisation) or to reduce cigarette consumption by at least 50% of baseline levels (cohort B only)
Time to smoking resumption | Month 6, Month 12, Month 24, Month 36, Month 48, Month 60 after randomization
  Evaluation of the time to smoking resumption (i;e; delay between randomization and smoking resumption) for the patients unable to achieve abstinence in the 2 arms (cohort B only)
Health-related quality of life | Month 6, Month 12 after randomization
  Evaluation of the health-related quality of life using quality of life questionnaire QLQ-C30 assessment (cohort B only)
Health-related quality of life | Month 6, Month 12 after randomization
  Evaluation of the health-related quality of life using quality of life questionnaire QLQ-H&N35 assessment (cohort B only)
Patients' preference to the 2 smoking cessation programs | Month 12 after randomization
  Evaluation of the patients' preference by assessement of the rate of patients who refuse the intensive and sustained smoking cessation program.

OTHER OUTCOMES:
Cost of the cessation program | Month 12 (M12) after randomization
  Cost of the cessation programs (Cohort B only): addictologist visits, nicotine replacement therapy, behaviorial and cognitive thérapies, psychological interventions...
Correlation between LOH status and smoking cessation | Month 6 and month 12 (M6, M12) after randomization
  - To analyze the LOH status at baseline (normal mucosa on resected specimen and tumor) and the dynamics of LOH changes in oral brushes (baseline, M6 and M12) to evaluate whether they may serve as a surrogate of smoking cessation (Cohort B only)
Prevalence of a panel of constitutional genomic variants in genes known to be associated with nicotine dependance | Day 0 (at randomization)
  Prevalence of a panel of constitutional genomic variants in genes known to be associated with nicotine dependance in patients refusing assistance for smoking cessation in comparison with patients willing to quit (Cohort B only)
Psychological evaluation | Within 2 months after randomization
  to determine psychological characteristics of patients, with a focus on patients who refuse assistance for smoking cessation in comparison with patients willing to quit, to decipher reasons for acceptance or refusal to enter an intensive smoking cessation program and to identify patients representations for their smoking/alcohol addiction and how patients understand their level of risk and cope/react with it (Cohort B only)
Sociological evaluation | After randomization and Month 6 after randomization
  to determine sociological characteristics of patients, with a focus on patients who refuse assistance for smoking cessation in comparison with patients willing to quit, to decipher reasons for acceptance or refusal to enter an intensive smoking cessation program and to identify patients representations for their smoking/alcohol addiction and how patients understand their level of risk and cope/react with it (Cohort B only)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SAINTIGNY, Dr, Principal Investigator — Centre Léon Bérard, Lyon, France
Locations (10):
- France (10):
  - Centre Hospitalier Annecy genevois, Annecy
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Centre Léon Bérard, Lyon
  - CHU de Montpellier, Hôpital Gui De Chauliac, Montpellier
  - AP-HP, Hôpital de la Pitié Salpêtrière, Paris
  - Hospices Civils de Lyon, Hôpital Lyon Sud, Pierre-Bénite
  - CHU de Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440